CLINICAL TRIAL: NCT01572454
Title: The Comparison of Serum Potassium Concentration, Antiarrhythmic Effect, and Myocardial Protective Effect Between Dexmedetomidine and Remifentanil Infusion in Patients Undergoing Coronary Artery Bypass Surgery
Brief Title: Comparison of Dexmedetomidine and Remifentanil Infusion During CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyun Sung Cho, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2012-02-012-001
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Coronary Artery Bypass Graft; Hypokalemia; Cardiac Arrhythmia; Dexmedetomidine; Remifentanil
Keywords: coronary artery bypass graft; hypokalemia; cardiac arrhythmia; dexmedetomidine; remifentanil
MeSH Terms: conditions — Hypokalemia; Arrhythmias, Cardiac | interventions — Dexmedetomidine; Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine group (Experimental): Dexmedetomidine infusion 0.2 mcg/kg/hr during anesthetic induction 0.3 - 0.7 mcg/kg/hr during the surgery
  Interventions: Drug: Dexmedetomidine infusion
- Remifentanil group (Active Comparator): Remifentanil infusion 0.05 - 0.3 mcg/kg/min during the anesthetic induction and surgery
  Interventions: Drug: Remifentanil infusion

INTERVENTIONS:
Drug: Dexmedetomidine infusion — Dexmedetomidine infusion 0.2 mcg/kg/hr during anesthetic induction 0.3 - 0.7 mcg/kg/hr during the surgery
  Other Names: Dexmedetomidine
  Arms: Dexmedetomidine group
Drug: Remifentanil infusion — Remifentanil infusion 0.05 - 0.3 mcg/kg/min during the anesthetic induction and surgery
  Other Names: Remifentanil
  Arms: Remifentanil group

SUMMARY:
We are trying to investigate whether intraoperative dexmedetomidine infusion could decrease the incidence of intraoperative hypokalemia and arrhythmia, and myocardial injury in patients undergoing off-pump coronary artery bypass graft, and trying compare these effects with those of remifentanil infusion.

DETAILED DESCRIPTION:
Alpha2-adrenergic agonist, dexmedetomidine, is recently used for sedation, analgesia or adjuvant to general anesthesia. Postsynaptic activation of alpha2 adrenoceptors in the central nervous system (CNS) inhibits sympathetic activity and thus can decrease blood pressure and heart rate. The blockade of sympathetic activity decrease the neuroendocrine stress response and may decrease the incidence of hypokalemia. The hypokalemia can increase the incidence of arrythmia, especially in cardiac patients. We postulated that dexmedetomidine could decrease the neuroendocrine stress response, thus decrease arrhythmia during cardiac surgery. Furthermore, dexmedetomidine have been reported to have cardioprotective effect with previous animal studies.

Therefore, the aim of the present study is to investigate whether the intraoperative dexmedetomidine infusion can reduce the incidence of hypokalemia and arrythmia, and myocardial injury in subjects undergoing off-pump coronary artery bypass graft. We are also trying to compare these effects with those of remifentanil infusion.

ELIGIBILITY:
Inclusion Criteria:

* Those undergoing off-pump coronary artery bypass graft during March, 2012 ~ February, 2013 in Samsung Medical Center
* Age between 20 and 70 yrs old

Exclusion Criteria:

* Any patients with plasma aldosterone, or glucocorticoid disorder including primary hyperaldosteronism, renovascular hypertension, rennin-secreting tumor, salt-wasting renal disease, Cushing syndrome
* Patients with recent exogenous steroid administration or previous diuretics therapy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
serum potassium concentration | at 24 hour before anesthetic induction
  serum potassium concentration at the day before anesthetic induction
serum potassium concentration | 1 minutes before anesthetic induction
  1 minutes before anesthetic induction (etomidate injection)
serum potassium concentration | 20 minutes after start of anesthetic induction
  serum potassium concentration 20 minutes after start of anesthetic induction (at the end of anesthetic induction)
serum potassium concentration | 2 hour after the start of anesthetic induction
  serum potassium concentration at 2 hour after anesthetic induction (after mammary artery dissection and graft formation)
serum potassium concentration | 3 hour after start of anesthetic induction
  serum potassium concentration at 3 hour after end of anesthetic induction (after the anastomosis of coronary graft)

SECONDARY OUTCOMES:
arterial blood gas analysis results | 24 hour, 1 min before anesthetic induction, 20 min, 2 and 3 hour after the start of anesthetic induction
  arterial blood gas analysis results
incidence of hypokalemia | 24 hour, 1 min before anesthetic induction, 20 min, 2 and 3 hour after the start of anesthetic induction
  incidence of hypokalemia (serum K < 3.5) incidence of hypokalemia (serum K < 4.5)
hemodynamic parameters | 24 hour, 1 min before anesthetic induction, 20 min, 2 and 3 hour after the start of anesthetic induction
  hemodynamic parameters (blood pressure, heart rate, central venous pressure, cardiac output, SvO2)
inotropics, vasopressor requirement | 24 hour, 1 min before anesthetic induction, 20 min, 2 and 3 hour after the start of anesthetic induction
  inotropics, vasopressor requirement
Myocardial injury marker | 2, 24, 48 hour after the end of surgery
  serum concentration of CK-MB, Troponin (i)as a marker for myocaridial injury
Left ventricular function | 72 hour before, during (immediate after grafting), 72 hour after surgery
  left ventricular function determined by Tei index, ejection fraction of preoperative, intraoperative, postoperative echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Sung Cho, MD, PhD, Principal Investigator — Samsung Medical Center; Won Ho Kim, MD, Principal Investigator — Samsung Medical Center; Young Tak Lee, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea